CLINICAL TRIAL: NCT00004831
Title: Study of Cysteine Hydrochloride for Erythropoietic Protoporphyria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: St. Luke's-Roosevelt Hospital Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13413; BWH-FDR000996-EF; SLRH-CU-FDR000996-EF
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1998-08

CONDITIONS: Erythropoietic Protoporphyria
Keywords: erythropoietic protoporphyria; inborn errors of metabolism; porphyria; rare disease
MeSH Terms: conditions — Protoporphyria, Erythropoietic; Metabolism, Inborn Errors; Porphyrias; Rare Diseases | interventions — Cysteine

INTERVENTIONS:
Drug: cysteine hydrochloride

SUMMARY:
OBJECTIVES:

I. Determine the efficacy of cysteine hydrochloride in preventing or decreasing photosensitivity in patients with erythropoietic protoporphyria.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled, crossover study.

Patients are randomly assigned to 1 of 2 groups to receive cysteine hydrochloride orally twice daily, 2 capsules with breakfast and 2 with lunch. Group 1 receives cysteine hydrochloride in drug ingestion period 1 followed by placebo in period 2. Group 2 receives placebo in period 1 followed by cysteine hydrochloride in period 2. Both groups ingest placebo for 1 week between the periods. Each drug ingestion period lasts 8 weeks.

Follow up phone calls are made at the end of months 1 and 3. All patients schedule follow up visits at the end of each drug ingestion period.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Documented erythropoietic protoporphyria Determination of elevated protoporphyrin within the past year Experiencing photosensitivity --Prior/Concurrent Therapy-- No concurrent use of betacarotene --Patient Characteristics-- Other: Not pregnant or nursing Fertile female patients must use effective contraception while on study and for 3 weeks thereafter

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 1996-10; Study Completion 1998-07

CONTACTS AND LOCATIONS:
Overall Officials: Micheline M Mathews-Roth, Study Chair — St. Luke's-Roosevelt Hospital Center